CLINICAL TRIAL: NCT01156558
Title: Early Outcome Assessment of Revision Total Knee Arthroplasty Using Metaphyseal Sleeves
Status: Completed | Type: Observational
Sponsor: Rothman Institute Orthopaedics (Other)
Collaborators: DePuy Orthopaedics (Industry)
Responsible Party: Matthew Austin, MD, Rothman Institute
Other Study IDs: 10FA01
Record Dates: First submitted 2010-07-01; First posted 2010-07-05 (Estimated); Last update posted 2011-03-31 (Estimated); Status verified 2011-03

CONDITIONS: Revision Total Knee Replacement

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Metaphyseal sleeves, through their design, could allow reconstruction of the knee in cases of severe bone loss by allowing rigid internal fixation and proper alignment of the extremity and components.

ELIGIBILITY:
Inclusion Criteria:

1. Revision knees with bone defect for which metaphyseal sleeve in femoral and/or tibial side is used
2. Cases with at least 2 year follow-up
3. Cases with regular follow-up visits completed

Exclusion Criteria:

1. Cemented sleeves
2. Patients with less than two year follow-up completed
3. Cases lost to follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Sequential assessment of 100 patients who have received a revision knee surgery for which metaphyseal sleeve was used in femoral and/or tibial side starting August 2007. Patients must meet inclusion/exclusion criteria for enrollment.
Sampling Method: Non-Probability Sample
Dates: Start 2010-06; Primary Completion 2010-07 (Actual); Study Completion 2010-07 (Actual)

PRIMARY OUTCOMES:
Implant survivorship 2 years following revision TKA

SECONDARY OUTCOMES:
Knee Society Score
KOOS score
Radiographic assessment 1 and 2 years following revision surgery